CLINICAL TRIAL: NCT01288391
Title: An Open Non-randomised Dose Escalation Trial Investigating the Safety and Pharmacokinetics of Single Intravenous Administrations of NNC128-0000-2011 in Patients With Haemophilia A or B
Brief Title: Investigating Safety and Pharmacokinetics of 2 Different Single Doses of NNC128-0000-2011 in Haemophilia A or B Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7128-3840; 2010-021127-28 (EudraCT Number); U1111-1118-6995 (Other: WHO); JapicCTI-111455 (Registry Identifier: JAPIC)
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100 mcg/kg (Experimental)
  Interventions: Drug: NNC 0128-0000-2011
- 200 mcg/kg (Experimental)
  Interventions: Drug: NNC 0128-0000-2011

INTERVENTIONS:
Drug: NNC 0128-0000-2011 — Single dose of 100 mcg/kg NNC128-0000-2011 administered i.v. (intravenously)
  Arms: 100 mcg/kg
Drug: NNC 0128-0000-2011 — Single dose of 200 mcg/kg NNC128-0000-2011 administered i.v. (intravenously)
  Arms: 200 mcg/kg

SUMMARY:
This trial is conducted in Europe and Japan. The aim of this trial is to assess the safety and pharmacokinetics (the rate at which the body eliminates the trial drug) of single doses of NNC128-0000-2011, when administered i.v. (intravenously) to haemophilia patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with haemophilia A or B (with or without inhibitors and irrespective of severity) based on medical records
* Japan: A legally acceptable representative (LAR) is required for patients between 18 and 19 years
* Body weight less than or equal to 100.0 kg
* Body Mass Index (BMI) less than or equal to 30.0 kg/m^2

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products (including rFVIIa)
* Previous participation in this trial defined as administration of trial product
* The receipt of any investigational product within 30 days prior to trial start (screening)
* Congenital or acquired coagulation disorders other than haemophilia A or B
* Receipt of Immune Tolerance Induction (ITI) within the last 30 days prior to screening
* Any surgery within 30 days prior to screening
* Planned surgery within the trial period
* Platelet count below 50,000 platelets/mcL (based on medical records within the last 1 month or laboratory results at screening)
* Prothrombin time (PT) above 4 times Upper limit of normal (ULN) or International normalised ratio (INR) greater than 1.7
* Hepatic dysfunction or severe hepatic disease as evaluated by the investigator (trial physician)
* Renal dysfunction (dialysis) and/or creatinine levels more than or equal to 20% above upper normal limit (according to medical records or laboratory results at screening)
* Advanced atherosclerotic disease (defined as known history of ischemic heart disease, ischemic stroke, etc.)
* Any disease, condition, or medication which, according to the investigator's (trial physician) judgement, could imply a potential hazard to the patient or interfere with the trial participation or trial outcome
* Mental incapacity, unwillingness to cooperate, or a language barrier precluding adequate understanding and cooperation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) | from first trial product administration until 12 weeks after last trial product administration
Frequency of serious adverse events (SAEs) | from first trial product administration until 12 weeks after last trial product administration
Frequency of MESIs (Medical Event of Special Interest) | from first trial product administration until 12 weeks after last trial product administration

SECONDARY OUTCOMES:
Neutralising antibodies against FVIIa and/or N7-GP | from first trial product administration until 12 weeks after last trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Berlin, Germany
- Kitakyushu, Japan
- Madrid, Spain

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com